CLINICAL TRIAL: NCT07150403
Title: A Phase II, Open-label, Non-comparative, Randomized Study of Second-line Doublet Chemotherapy (FOLFOX or FOLFIRI) Plus Fruquintinib Versus Doublet Chemotherapy (FOLFOX or FOLFIRI) Plus Bevacizumab in Metastatic Colorectal Cancer
Brief Title: Second-line Doublet Chemotherapy (FOLFOX or FOLFIRI) Plus Fruquintinib Versus Doublet Chemotherapy (FOLFOX or FOLFIRI) Plus Bevacizumab in Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 115 - FFCD 2406-ULYSSE; 2025-522108-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Carcinoma (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Irinotecan; HMPL-013; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm A FOLFOX/FOLFIRI + Fruquintinib (Experimental): FOLFOX (if FOLFIRI in first line) OR FOLFIRI (if FOLFOX in first line); D1 = D15 + FRUQUINTINIB
  Interventions: Drug: Oxaliplatin intravenous; Drug: 5 FU bolus; Drug: Folinic acid; Drug: 5 FU continuous; Drug: Irinotecan; Drug: FRUQUINTINIB
- Control arm B FOLFOX/FOLFIRI + Bevacizumab (Active Comparator): FOLFOX (if FOLFIRI in first line) OR FOLFIRI (if FOLFOX in first line); D1 = D15 + BEVACIZUMAB (D1 = D15)
  Interventions: Drug: Oxaliplatin intravenous; Drug: 5 FU bolus; Drug: Folinic acid; Drug: 5 FU continuous; Drug: Irinotecan; Drug: BEVACIZUMAB

INTERVENTIONS:
Drug: Oxaliplatin intravenous — 85 mg/m² IV over 2 hours ; 1 cycle each 15 days
Drug: 5 FU bolus — 5 fluorouracil : 400 mg/m² in bolus of 10 minutes (intravenous)
Drug: Folinic acid — 400 mg/m² in intravenous
Drug: 5 FU continuous — 2400 mg/m² intravenously over 46 hours
Drug: Irinotecan — 180 mg/m² IV over 1h30
Drug: FRUQUINTINIB — 5 mg capsule, taken orally, once daily for 3 weeks, followed by a 7-day break, then resumed (Day 1= Day 29).
  Arms: Experimental arm A FOLFOX/FOLFIRI + Fruquintinib
Drug: BEVACIZUMAB — 5 mg/kg over 90 minutes for the 1st course and in case of good tolerance the 2nd course should be administered over 60 minutes. The next courses should be administered in 30 minutes in case of good tolerance during the 2nd course
  Arms: Control arm B FOLFOX/FOLFIRI + Bevacizumab

SUMMARY:
The standard second-line treatment for metastatic colorectal cancer (mCRC) involves chemotherapy (FOLFOX or FOLFIRI) combined with an antiangiogenic agent, such as bevacizumab or aflibercept. Maintaining VEGF inhibition between first and second-line treatments has shown modest clinical benefits, with exploratory analyses suggesting that bevacizumab is more effective in smaller tumors. The ULYSSE trial aims to evaluate the efficacy and safety of Fruquintinib, a potent antiangiogenic agent, combined with a doublet chemotherapy (FOLFOX or FOLFIRI) in second-line treatment for BRAF wild-type, MSS mCRC patients who have failed prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years and ≤ 80 years; provided the score of the G8 geriatric questionnaire is >14 for patients 75 years or older
* Patients with a histologically confirmed diagnosis of metastatic colorectal cancer (mCRC), with a documented disease progression (as per RECIST v1.1, assessed by the investigator and confirmed through CT or MRI).
* Patients must have previously received first-line therapy with Bevacizumab or an EGFRi, in combination with either FOLFOX or FOLFIRI, for non-resectable mCRC. Patients who progressed during the adjuvant chemotherapy (FOLFOX) or within the 6 months following its completion are eligible for inclusion
* Patients must have an unresectable tumor at the time of enrollment.
* Patients must have at least one measurable/evaluable metastatic lesion according to RECIST v1.1 criteria; images have to be available for collection
* Metastases not amenable to surgery and/or thermo-ablation and/or stereotaxic radiotherapy
* WHO performance status 0 or 1
* Available parameters to compute the SPOD score: WHO PS, hemoglobin, platelet count, WBC/absolute neutrophil count ratio, lactate dehydrogenase (LDH), alkaline phosphatase, and the number of metastatic sites.
* Adequate liver functions: Total Bilirubinemia < 2,5 ULN, AST and ALT ≤ 5 ULN
* Adequate hematological (Hemoglobin ≥10g/dL, platelets ≥100G/L, neutrophils ≥1.5G/L) and renal (creatinine clearance ≥ 50 mL/min according to CKD-EPI) functions
* Proteinuria < 2+ (dipstick urinalysis) (if 2+ or more, proteinuria must be ≤1g/24hour)
* Life expectancy ≥ 3 months
* Women of childbearing potential must agree to use a highly effective method of contraception during the trial and for at least 15 months after discontinuation of the experimental treatments. Men who have sexual relations with women of childbearing potential must agree to use contraception during treatment and for at least 12 months after discontinuation of the experimental treatments
* Ability of the patient to understand, sign and date the information note and informed consent form before any study specific procedures
* Patient affiliated to a social security scheme
* Available tumor sample and pathology report for collection

Exclusion Criteria:

* - Patients who have received more than one prior systemic therapy
* FOLFIRINOX Regimen +/- targeted therapy in the first line setting
* Unknown RAS status
* BRAF V600E mutated tumor
* MSI/dMMR tumor
* Known brain metastasis
* Known peritoneal carcinomatosis if there are signs of clinical occlusion or sub-occlusion
* History of gastric ulceration, or myocardial infarction, or severe coronaropathy or severe cardiac dysfunction, within the past 6 months prior to treatment start
* Patients with dihydropyrimidine dehydrogenase deficiency (uracilemia ≥ 16 ng/mL)
* Hypersensitivity to one of the study drugs or one of its excipients
* Inability to swallow capsules
* Live attenuated vaccines 30 days prior to treatment start
* Untreated bone fracture
* Significant haemorrhagic diathesis or coagulopathy (in the absence of anti-coagulant treatment)
* Major surgery, open biopsy or major traumatic lesion in the prior 30 days or the need for major surgery during the trial
* Pregnant or breastfeeding woman or patients with no adequate contraception
* Known Uridine Diphosphate Glucuronyltransferase (UGT1A1) deficiency or known Gilbert disease
* Strong inducers of CYP3A4 (treatment with St John's Wort (Hypericum perforatum), fampicin, phenobarbital, primidone, phenytoin and carbamazepine)

  -- Strong inhibitors of CYP3A4, continuous use of azole antifungals (posaconazole, voriconazole, itraconazole, isavuconazole), ritonavir, verapamil, diltiazem, grapefruit juice (equivalent to half a fresh grapefruit/day)
* Concomitant or recent treatment with sorivudine or its analogs (including brivudine) within 4 weeks prior to the administration of protocol treatment (related to Fluorouracil)
* Concomitant treatment with phenytoin or its analogs
* QT/QTc interval > 450 ms for men and > 470 ms for women
* Uncontrolled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg) or history of hypertensive crisis (TA systolic> 20 mmHg) or hypertensive encephalopathy
* History of veinous thromboembolic events, including deep vein thrombosis and pulmonary embolism, within the past month prior to study enrollment
* History of stroke and/or transient ischemic attack (TIA) within the past 12 months
* Residual Oxaliplatin neuropathy (grade ≥ 2) counter indicates FOLFOX administration
* Persistence of clinically significant symptoms after a thromboembolic event despite anticoagulant treatment
* Arterial thromboembolism (myocardial infarction, stroke, transient ischemic attack) occurring under antiangiogenic therapy
* Other active cancers or history of cancer treated within the last 5 years except for carcinoma in situ of the cervix or basal cell or squamous cell skin carcinoma or any other carcinoma in situ, considered cured
* Persons deprived of liberty or under guardianship or unable of giving consent
* Inability to undergo the medical follow-up of the trial for geographical, social or psychological reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | at 4 months after the start of treatment
  the percentage of patients with a complete response, a partial response or a stable disease at 4 months after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (45):
- France (45):
  - ICO Site Paul Papin, Angers
  - Les Bonnettes, Arras
  - Ght Unyon Auxerre, Auxerre
  - Bayeux Ch, Bayeux
  - Cote Basque, Bayonne
  - Beauvais Ch, Beauvais
  - Jean Minjoz, Besançon
  - Centre Pierre Curie, Beuvry
  - BERGONIÉ, Bordeaux
  - TIVOLI, Bordeaux
  - Chauny Ch, Chauny
  - Cholet Ch, Cholet
  - Saint Côme, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - GHPSO Site de Creil, Creil
  - Centre Leonard de Vinci, Dechy
  - Dijon Bourgogne, Dijon
  - Institut de cancérologie de Bourgogne GRReCC, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Docteur Schaffner, Lens
  - Franco Britannique, Levallois-Perret
  - Jean Mermoz, Lyon
  - La Timone, Marseille
  - LAYNÉ CH, Mont-de-Marsan
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Confluent Sas, Nantes
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Européen G Pompidou, Paris
  - La Pitié Salpêtrière, Paris
  - Saint Louis, Paris
  - La Miletrie, Poitiers
  - Jean Godinot, Reims
  - Robert Debré, Reims
  - Saint Gregoire Chp, Saint-Grégoire
  - ICO Site René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de L'Estuaire, Saint-Nazaire
  - Hopital Nord Chu Saint Etienne, Saint-Priest-en-Jarez
  - Saint Malo Ch, St-Malo
  - ICAN Institut de Cancérologie de Strasbourg Europe, Strasbourg
  - Sainte Anne, Strasbourg
  - LEMAN, Thonon-les-Bains
  - Valence Ch, Valence
  - BRABOIS, Vandœuvre-lès-Nancy
  - Ch Nord Ouest, Villefranche-sur-Saône
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No